# **Document Coversheet**

Study Title: Responses of Adults Smoking Nondaily and Daily in the Experimental Tobacco Marketplace

| Institution/Site: | University of Kentucky |
|----------------------------------|------------------------|
| Document (Approval/Update) Date: | 8/18/23 |
| NCT Number: | NCT06988371 |
| IRB Number | 99596 |
| Coversheet created: | 9/16/2025 |

## University of Kentucky Consent to Participate in Research

Research Title: Modeling Tobacco Regulatory Impacts Among Adults Smoking Nondaily and Daily Using the

Experimental Tobacco Marketplace

Protocol #: 99596

Researcher: Bethany Shorey Fennell, PhD, Department of Family & Community Medicine, University of Kentucky

Contact Information: phone: (859) 562-2714, email: bethany.shoreyfennell@uky.edu

## Purpose, Procedure, and Duration:

We are researchers from the University of Kentucky inviting you to participate in a survey. We want to learn more the potential impact of tobacco regulations that could affect the availability of tobacco products.

If you agree to participate in our study, you will be asked to complete an online survey that will ask about your behavior and health in the last three months. The survey will take about approximately 40 minutes to complete.

# **Eligibility:**

You must meet the following requirements to participate in this research study:

- Be at least 18 years of age
- Speak and understand English
- Live in the United States
- Use cigarettes 4-30 days in the past 30 days

#### **Benefits:**

You may not benefit personally from being in this study, but your answers could help us learn about the potential impact of proposed tobacco product regulations in your community.

#### Risks:

Participants in this study will be asked to share potentially personal information about their tobacco and other substance use. Some of our questions may make you feel uncomfortable or upset. You can stop the survey at any time.

We have contacted you through Prolific, a market research panel aggregator, to collect your responses. They may have Terms of Service and Privacy policies outside of the control of the University of Kentucky that allows them to use your data for other purposes.

We will make every effort to safeguard your data. However, we cannot guarantee the security of data obtained via the internet.

#### Reward:

Upon completion of the study, you will be redirected to Prolific and receive compensation in the amount of \$12.00.

## **Alternative Opportunities:**

We know of no alternative except not to participate in our study. If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits or rights you would normally have if you choose not to volunteer.

ORI F1.0370 Rev 6/21/2023 Rev 8/18/2023

# **Privacy and Future Use:**

Your responses to the research survey are anonymous. That means we won't know which responses are yours. We won't collect names, internet addresses, email addresses, or any other identifiable information and Prolific keeps this information confidential from researchers.

We may use your responses in future research or share them with other researchers.

## **Complaints or Concerns:**

If you have questions about the study, please contact the researcher using the contact information provided above.

If you have complaints or concerns about your rights as a research volunteer, you can contact the staff in the University of Kentucky Office of Research Integrity at 859-257-9428 or toll-free at 1-866-400-9428.

Thank you for taking the time to consider our study. You do not have to participate in our study, but we hope you will.

Please select an option below to indicate you read this information and you wish to take the survey:

- 1. I agree to be in this study
- 2. I don't want to be in this study

Check "Request for Waiver of Signature" in the Informed Consent section of your protocol application if you use this template for anonymous research.